CLINICAL TRIAL: NCT00168935
Title: Malnutrition in Gastroenterology Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Prof Herbert Lochs, Charite University Medicine
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AN1
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2005-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

INTERVENTIONS:
Drug: Fresubin protein energy Drink (CAVE! nutritional intervention)

SUMMARY:
Background: Malnutrition is frequently occurring in sick patients and is associated with a higher morbidity and mortality. Muscle dysfunction is a common finding in malnutrition which leads to a reduced functional status and quality of life.

Specific aims: The purpose of the study is to evaluate the effect of a three month nutritional intervention with oral supplements on nutritional status, muscle function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Malnutrition
* Benign disease

Exclusion Criteria:

* Malignant disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-03; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Pirlich, MD, Principal Investigator — Charite Universitätsmedizin Berlin ,Klinik für Gastroenterologie CCM
Locations (1):
- Charite Universitätsmedizin Berlin CCm, Berlin, Germany

REFERENCES:
- [Derived] Norman K, Pirlich M, Smoliner C, Kilbert A, Schulzke JD, Ockenga J, Lochs H, Reinhold T. Cost-effectiveness of a 3-month intervention with oral nutritional supplements in disease-related malnutrition: a randomised controlled pilot study. Eur J Clin Nutr. 2011 Jun;65(6):735-42. doi: 10.1038/ejcn.2011.31. Epub 2011 Mar 16. PMID 21407248